CLINICAL TRIAL: NCT05366231
Title: A Randomized, Open-label, Positive Drug Parallel Controlled Clinical Trial of Kesuting Syrup in the Treatment of COVID-19 (Light)
Brief Title: Kesuting Syrup in the Treatment of Corona Virus Disease 2019 (COVID-19)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guizhou Bailing Group Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KST-22-01
Record Dates: First submitted 2022-04-28; First posted 2022-05-09 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pneumonia; Cough
Keywords: Kesuting syrup; COVID-19
MeSH Terms: conditions — Cough; COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kesuting syrup group (Experimental): Kesuting syrup, the tested drug of this study.
  Interventions: Drug: Kesuting syrup
- LianHuaQingWen Granules Control group (Active Comparator): LianHuaQingWen Granules, referring to "Diagnosis and Treatment Protocol for COVID-19 (Trial Version 9)", a NMPA approved drug for light and common patients with novel coronavirus during medical observation and clinical treatment,is adopted as active comparator in this study.
  Interventions: Drug: LianHuaQingWen Granules

INTERVENTIONS:
Drug: Kesuting syrup — Conventional treatment + Kesuting Syrup, take orally, 20 ml once, three times a day.Conventional treatment refer to "Diagnosis and Treatment Protocol for COVID-19 (Trial Version 9 or later)". Except for the test drugs, during the observation period, it is prohibited to use other Chinese and Western medicines for cough and phlegm elimination for treatment. If combined use is required, it shall be recorded truthfully.
  Other Names: Kesuting Tangjiang
  Arms: Kesuting syrup group
Drug: LianHuaQingWen Granules — Conventional treatment + LianHuaQingWen Granules, orally, 1 bag at a time, 3 times a day.Conventional treatment refer to "Diagnosis and Treatment Protocol for COVID-19 (Trial Version 9 or later)".Except for the test drugs, during the observation period, it is prohibited to use other Chinese and Western medicines for cough and phlegm elimination for treatment. If combined use is required, it shall be recorded truthfully.
  Other Names: Lianhua Qingwen Keli
  Arms: LianHuaQingWen Granules Control group

SUMMARY:
This trial is an exploratory study, aiming to explore the preliminary efficacy and safety of Kesuting Syrup in the treatment of novel coronavirus pneumonia. It is planned to include a total of 200 cases. Kesuting Syrup test group: Lianhua Qingwen Granules control group = 1:1, each 100 cases in each group.

DETAILED DESCRIPTION:
This trial is a randomized, open-label, parallel-controlled clinical trial of active drugs.With reference to"Diagnosis and Treatment Protocol for COVID-19(Trial Version 9)", Lianhua Qingwen Granules have been recommended for mild and common patients during the medical observation period and clinical treatment period of the new coronavirus. The purpose of the experiment is preliminary evaluate the clinical efficacy and safety of Kesuting syrup in the treatment of COVID-19 (Light) .

ELIGIBILITY:
Inclusion Criteria:

1. Persons with COVID-19 (Light) in accordance with the "Diagnosis and Treatment Protocol for COVID-19 (Trial Version 9 or later)" .
2. Subjects with cough score > 1.
3. Inpatients aged 18 ≤ age ≤ 75 years old, regardless of gender.
4. Subjects (including male subjects) who have no plans for pregnancy, sperm donation, or egg donation in the past six months, and who are willing to take effective contraceptive measures from the first dose to 3 months after the last dose.
5. Subjects fully understand the purpose, nature, content, process and possible adverse reactions of the trial, and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Ordinary, severe, and critically ill patients with novel coronavirus pneumonia, or patients with novel coronavirus pneumonia requiring mechanical ventilation.
2. patients with asthma attack, suppurative tonsillitis, acute and chronic bronchitis, sinusitis, otitis media and other respiratory diseases that affect clinical trial evaluation; And chest CT confirmed the existence of severe pulmonary interstitial lesions, bronchiectasis, obstructive pulmonary disease and other basic pulmonary diseases.
3. Patients with respiratory tract infections caused by basic diseases such as primary immunodeficiency disease, acquired immunodeficiency syndrome, congenital respiratory malformation, congenital heart disease, gastroesophageal reflux disease, and abnormal lung development.
4. According to the judgment of the investigator, past or current chronic or serious diseases may affect participation in the trial or the outcome of the study, including but not limited to gastrointestinal system, cardiovascular and cerebrovascular system, liver, kidney, hematopoietic system, lymphatic system Patients with diseases of the system, endocrine system, immune system, malignant tumor, severe malnutrition, nervous system and endocrine system,as well as those currently suffering from human immunodeficiency virus (HIV) infection, splenectomy, organ transplantation and other diseases that seriously affect the immune system.
5. Those who cannot cooperate in mental state, those who suffer from mental illness, cannot control themselves, and cannot express themselves clearly.
6. Patients with diabetes.
7. Patients with poorly controlled hypertension: low pressure ≥110 mmHg or high pressure ≥180 mmHg.
8. Alanine Aminotransterase（ALT）and Aspartate Aminotransferase（AST） ≥ 1.5 times the upper limit of normal, and Scr > the upper limit of normal.
9. Those who have a history of specific allergies (such as asthma, measles, eczema, etc.), or allergic constitution (such as those who are allergic to two or more drugs, foods such as milk and pollen), or are allergic to the drug ingredients of Kesuting Syrup and Lianhua Qingwen Granules.
10. Those with a history of drug abuse or dependence within 6 months before randomization.
11. Those who have used any Chinese and Western medicines to relieve cough and reduce phlegm within 24 hours before randomization.
12. Pregnant and lactating female patients.
13. Patients who have participated in or are participating in clinical trials of other drugs within 3 months prior to screening.
14. Investigators deem others unsuitable to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-05-08 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Cough efficacy assessed by cough symptom scale（CSS） | at baseline
  Recording and evaluation of cough symptom scores by CSS(evaluation standards on the basis of the diagnosis and treatment of coughing guide (2015)),included daytime and nighttime cough symptom assessments,0 for normal, 1 for mild, 2 for moderate and 3 for severe,scores added.
Cough efficacy by cough symptom scale（CSS） | at 7 days of medication
  Recording and evaluation of cough symptom scores by CSS(evaluation standards on the basis of the diagnosis and treatment of coughing guide (2015)),included daytime and nighttime cough symptom assessments,0 for normal, 1 for mild, 2 for moderate and 3 for severe,scores added.
Cough efficacy by cough symptom scale（CSS） | up to 14 days
  Recording and evaluation of cough symptom scores by CSS(evaluation standards on the basis of the diagnosis and treatment of coughing guide (2015)),included daytime and nighttime cough symptom assessments,0 for normal, 1 for mild, 2 for moderate and 3 for severe,scores added.
Cough disappearance time | Baseline, at cough disappears up to 14 days
  Change from Baseline，record the time in hour it takes for the cough to go away .

SECONDARY OUTCOMES:
Disease recovery time | up to 14 days
  Evaluation of treatment endpoints
Disease recovery rate | up to 14 days
  Evaluation of treatment endpoints
The time of negative conversion of new coronavirus. | at baseline, 7 days of medication, up to 14 days
  Record the time of negative conversion of new coronavirus.
The rate of negative conversion of new coronavirus. | at baseline, 7 days of medication, up to 14 days
  Record rate of negative conversion of new coronavirus.
Efficacy of fever assessed by the single symptom grading standard formulated | at baseline, 7 days of medication,up to 14 days
  Change from baseline individual symptoms (fever）markedly effective, effective or ineffective)at 7 days of medication and end of treatment,up to 14 days,according to the single symptom grading standard formulated.
Efficacy of fatigue assessed by the single symptom grading standard formulated | at baseline, 7 days of medication,up to 14 days
  Change from baseline individual symptoms (fatigue）markedly effective, effective or ineffective)at 7 days of medication and end of treatment,up to 14 days,according to the single symptom grading standard formulated.
Efficacy of sore throat assessed by the single symptom grading standard formulated | at baseline, 7 days of medication,up to 14 days
  Change from baseline individual symptoms ( sore throat)markedly effective, effective or ineffective)at 7 days of medication and end of treatment,up to 14 days,according to the single symptom grading standard formulated.
Incidence of severe/critical illness | up to 14 days
  Assess the incidence of severe/critical illness

CONTACTS AND LOCATIONS:
Overall Officials: Yun Ling, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No